CLINICAL TRIAL: NCT05283304
Title: Randomized, Double-blind, Placebo-controlled Trial of Monthly Injectable Buprenorphine (BUP) for Methamphetamine (MA) Use Disorder
Brief Title: Monthly Injectable BUP for MA Use Disorder (MURB) Trial
Acronym: CTN-0110
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Side effects of medication
Sponsor: Madhukar H. Trivedi, MD (Other)
Responsible Party: Sponsor-Investigator, Madhukar H. Trivedi, MD, PROFESSOR, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA CTN Protocol 0110
Record Dates: First submitted 2022-02-28; First posted 2022-03-16 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Methamphetamine-dependence
MeSH Terms: interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the Data and Statistic Center (DSC) staff overseeing the random assignment schedule, a few Clinical Coordinating Center (CCC) staff, the central research pharmacy staff preparing the study medication and a single study staff role (Medical Personnel) to administer the injections are unblinded; all other study personnel and participants will remain blinded to treatment arm until the nationwide completion of the trial and the database is formally locked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Injectable Buprenorphine (BUP-inj) (Experimental): Following successful titration to 16 mg of daily sublingual buprenorphine, the participants will then transition to injectable buprenorphine (300 mg dose) every 4 weeks
  Interventions: Drug: Buprenorphine injection (BUP-Inj)
- Injectable Placebo (PBO-inj) (Placebo Comparator): Following successful titration to 16 mg of daily sublingual buprenorphine, the participants will then transition to injectable placebo (300 mg dose) every 4 weeks.
  Interventions: Other: Placebo injection

INTERVENTIONS:
Drug: Buprenorphine injection (BUP-Inj) — Sublingual Buprenorphine induction, then SublocadeTM, Indivior injectable (300mg)
  Other Names: SublocadeTM, Indivior
  Arms: Injectable Buprenorphine (BUP-inj)
Other: Placebo injection — Sublingual buprenorphine induction, then Placebo injectable (300 mg)
  Other Names: Placebo injection (PBO-Inj)
  Arms: Injectable Placebo (PBO-inj)

SUMMARY:
This study is a 12-week randomized, double-blind, placebo-controlled trial that will investigate the use of injectable buprenorphine (BUP-Inj) compared to injectable placebo (PBO-Inj) for the treatment of methamphetamine use disorder (MUD) among individuals with mild co-use of opioids.

DETAILED DESCRIPTION:
Primary Objective: To evaluate whether assignment to 12 weeks of outpatient BUP-Inj compared to 12 weeks of outpatient PBO-Inj reduces MA use (as measured by twice-weekly urine drug screens (UDS)) during Weeks 9-12 in participants with moderate to severe MUD with co-occurring mild opioid use disorder (OUD) or opioid misuse not warranting medication for opioid use disorder (MOUD).

Secondary Objectives: To evaluate whether assignment to 12 weeks of outpatient BUP-Inj compared to 12 weeks of outpatient PBO-Inj among participants with moderate to severe MUD with co-occurring mild OUD or opioid misuse not warranting MOUD improves: 1) outcomes related to alternate measures of MA use including total number of MA negative urine drug screens (UDS) during study and self-reported days of MA use; 2) measures of opioid use and self-reported frequency of opioid use; and 3) measures of MA and opioid co-use and self-reported days of MA and opioid co-use.

ELIGIBILITY:
Inclusion Criteria:

* Study participants must:

  1. Be 18 to 65 years of age, inclusive;
  2. Able to understand and speak English or Spanish
  3. Be interested in reducing or stopping MA use;
  4. Meet Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria for moderate or severe MUD (4 or more criteria);
  5. Self-report MA use on 18 or more days in the 30-day period prior to written consent using the TLFB;
  6. Provide at least 2 urine samples positive for MA out of a possible 3 tests to occur at clinic visits within a 10-day period with at least 2 days between visits;
  7. Meet DSM-5 criteria for mild OUD (at least 2 but no more than 3 criteria) prior to randomization OR opioid misuse demonstrated by self-report of opioid use of at least 2 days in the 30-day period prior to written consent using the TLFB;
  8. Provide a urine drug screen negative for opioids at least once during the screening period and on the day of expected randomization to indicate control over opioid use;
  9. Have a Clinical Opiate Withdrawal Scale (COWS) score of ≤8 at both a screening visit on which they provide a UDS negative for opioids and on the day of randomization.
  10. If female, agree to use acceptable methods of contraception and have periodic urine pregnancy testing during participation in the study unless unable to get pregnant;
  11. Be willing and able to provide consent and comply with all study procedures and medication instructions.

Exclusion Criteria:

* Study participants must not:

  1. Have suicidal or homicidal ideation that requires immediate attention;
  2. Have evidence of prolongation of the corrected QT interval (QTc) or any other finding on the screening ECG that, in the opinion of the Medical Clinician, would preclude safe participation in the study (e.g., hypokalemia, unstable atrial fibrillation) and be at significant risk for serious cardiac adverse events;
  3. Have a laboratory value with total bilirubin ≥1.5 × upper limit of normal (ULN), alanine aminotransferase (ALT) ≥3 × ULN, aspartate aminotransferase (AST) ≥5 × ULN, or serum creatinine >2 × ULN;
  4. Have been in a study of pharmacological or behavioral treatment for addiction within 6 months prior to written study consent (smoking cessation excepted);
  5. Have taken an investigational drug in another study within 30 days prior to written study consent;
  6. Have been prescribed and taken buprenorphine or methadone within 30 days prior to written study consent;
  7. Be concurrently enrolled in formal behavioral or pharmacological addiction treatment services at the time of written consent;
  8. Be receiving ongoing treatment of medications that are clinically relevant Cytochrome P450 3A4 (CYP 3A4) or Cytochrome P4502C8 (CYP 2C8) inducers or inhibitors (e.g., rifampicin, azole antifungals, macrolide antibiotics), Class IA antiarrhythmic medications (e.g., quinidine, procainamide, disopyramide) or Class III antiarrhythmic medications (e.g., sotalol, amiodarone) at the time of randomization that, in the judgment of the Medical Clinician, could interact adversely with study medications or put them at significant risk for development of serotonin syndrome;
  9. Have a current pattern of alcohol, benzodiazepine, or other sedative hypnotic use which would preclude safe participation in the study as determined by the Medical Clinician;
  10. Have a surgery planned or scheduled, or other treatment that would require the use of opioid-containing medications (e.g., opioid analgesics) during the study period;
  11. Currently or soon to be in jail or prison; currently in any inpatient overnight facility as required by court of law or have pending legal action or other situation that could prevent participation in the study or in any study activities;
  12. If biologically female, be currently pregnant, breastfeeding, or planning on conception;
  13. Hypersensitivity (e.g., anaphylaxis) to buprenorphine or any component of the ATRIGEL formulation or their excipients;
  14. Have an abdominal area unsuitable for subcutaneous injections by the judgment of the Medical Clinician;
  15. Have other medical, psychiatric or other factors that in the judgment of the Medical Clinician could make participation difficult or unsafe.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar Trivedi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (6):
- United States (6):
  - UCLA Vine Street Clinic, Los Angeles, California
  - Highland Hospital, Alameda Health System, Oakland, California
  - Oklahoma State University, Center for Health Sciences, Tulsa, Oklahoma
  - CODA, Portland, Oregon
  - UTSW Medical Center, Center for Depression Research and Clinical Care, Dallas, Texas
  - University of Washington Medicine-Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be available to researchers on the website https://datashare.nida.nih.gov/ after the study is complete and the data is analyzed. This website will not include information that can identify individual study participants. The following information will be posted: Study protocol, reference to study publication of primary outcome, data sets (SAS and ASCII ), annotated case report forms, define file (also known as Data Dictionary), study-specific de-identification notes. Prior to downloading any study data, the user will be prompted to complete a registration agreement for data use. Users will have to register a name and valid e-mail address in order to download data and to accept their responsibility for using data in accordance with the National Institute on Drug Abuse (NIDA) Data Share Agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the study is complete and the data is analyzed
Access Criteria: Study-specific de-identification notes will be posted on the website (URL provided here)
URL: https://datashare.nida.nih.gov/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 18 enrolled participants randomized, 2 withdrew prior to starting sublingual buprenorphine (SL-BUP) induction procedure and only the participants who successfully completed the open-label SL-BUP induction procedure started the Study Medication [injectable formulation (experimental/placebo)] as assigned in the table below.
Period: Overall Study
Arm/Group | Injectable Buprenorphine (BUP-inj) | Injectable Placebo (PBO-inj)
Started | 2 | 4
Completed | 1 | 4
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics collected for all the18 enrolled & randomized participants are reported here. 2 subjects withdrew consent prior to starting sublingual buprenorphine (SL-BUP) induction procedure and only the participants who successfully completed the open-label SL-BUP induction procedures started the study medication [injectable formulation (experimental/placebo)] that is reflected in Participant Flow module and that number is different from analysis population reported in this module.
Groups:
- Total: Total of all reporting groups
Arm/Group | Injectable Buprenorphine (BUP-inj) | Injectable Placebo (PBO-inj) | Total
Number analyzed (Participants) | 5 | 13 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 13 | 18
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 4 | 9 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 4 | 10 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 3 | 7 | 10
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Methamphetamine-negative Urine Samples
Description: Number of Methamphetamine (MA)-negative Urine Drug Screen (UDS) results obtained during Weeks 9 through 12 of the medication phase is measured for the BUP-Inj and PBO-Inj conditions. Number of UDS results / number of expected UDS results. Two UDS results were expected each week.
Time Frame: weeks 9-12
Measure: Count of Units; unit: urine samples
Units Other Than Participants: urine samples
Arm/Group | Injectable Buprenorphine (BUP-inj) | Injectable Placebo (PBO-inj)
Number analyzed (Participants) | 2 | 4
Number analyzed (urine samples) | 16 | 32
urine samples | 0 | 0

2. Secondary Outcome: Treatment Effective Score (TES) for MA-negative UDS Results
Description: The TES is defined to be the number of MA negative UDS divided by the number of possible UDS collected during the study. In this study there are 24 possible UDS collections so the number of MA negative UDS is divided by 24. Possible score ranges from 0-24; with higher score indicating better outcome.
Time Frame: weeks 1-12
Measure: Median (Inter-Quartile Range); unit: score on a scale
Units Other Than Participants: urine samples
Arm/Group | Injectable Buprenorphine (BUP-inj) | Injectable Placebo (PBO-inj)
Number analyzed (Participants) | 2 | 4
Number analyzed (urine samples) | 48 | 96
score on a scale | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Number of Days of Methamphetamine Use During the Medication Phase
Description: Number of days of methamphetamine use during treatment will be measured using Timeline Followback (TLFB) procedure which will be administered to document the participant's self-reported use during Weeks 1-12. Possible scores range from 0-84, with lower scores indicating better outcome.
Time Frame: weeks 1-12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Injectable Buprenorphine (BUP-inj) | Injectable Placebo (PBO-inj)
Number analyzed (Participants) | 2 | 4
days | 56.0 (25.46) | 53.8 (27.54)

4. Secondary Outcome: Treatment Effective Score (TES) for Opioid Negative UDS Results
Description: The TES is defined to be the number of UDS results negative for opioids divided by the number of possible UDS collected during the study. In this study there are 24 possible UDS collections, so the number of opioid negative UDS is divided by 24. Possible score ranges from 0-24; with higher score indicating better outcome.
Time Frame: weeks 1-12
Measure: Median (Inter-Quartile Range); unit: score on a scale
Units Other Than Participants: urine samples
Arm/Group | Injectable Buprenorphine (BUP-inj) | Injectable Placebo (PBO-inj)
Number analyzed (Participants) | 2 | 4
Number analyzed (urine samples) | 48 | 96
score on a scale | 0.62 [0.5 to 0.75] | 0.75 [0.48 to 0.9]

5. Secondary Outcome: Number of Days of Opioid Use During the Medication Phase
Description: Number of days of opioid use during treatment will be measured using Timeline Followback (TLFB) procedure which will be administered to document the participant's self-reported opioid use at week 12. Possible scores range from 0-84, with lower scores indicating better outcome.
Time Frame: weeks 1-12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Injectable Buprenorphine (BUP-inj) | Injectable Placebo (PBO-inj)
Number analyzed (Participants) | 2 | 4
days | 0 (0) | 0 (0)

6. Secondary Outcome: Treatment Effective Score (TES) for MA and Opioid Co-Use Compiled
Description: The TES is defined to be the number of MA and Opioid Co-Use negative UDS divided by the number of possible UDS collected during the study. In this study there are 24 possible UDS collections, so the number of MA and Opioid Co-Use negative UDS is divided by 24. Possible score ranges from 0-24; with higher score indicating better outcome.
Time Frame: weeks 1-12
Measure: Median (Inter-Quartile Range); unit: score on a scale
Units Other Than Participants: urine samples
Arm/Group | Injectable Buprenorphine (BUP-inj) | Injectable Placebo (PBO-inj)
Number analyzed (Participants) | 2 | 4
Number analyzed (urine samples) | 48 | 96
score on a scale | 0 [0 to 0] | 0 [0 to 0]

7. Secondary Outcome: Number of Days of MA and Opioid Co-use During the Medication Phase
Description: Number of days of MA and opioid co-use during treatment will be measured using Timeline Followback (TLFB) procedure which will be administered to document the participant's self-reported use of substances for each day at week 12. Possible scores range from 0-84, with lower scores indicating better outcome.
Time Frame: weeks 1-12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Injectable Buprenorphine (BUP-inj) | Injectable Placebo (PBO-inj)
Number analyzed (Participants) | 2 | 4
days | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: Adverse event assessment will initiate with participant written informed consent to 30 days post last study visit (approximately 19 weeks).
Description: All Adverse events that occurred during the sublingual buprenorphine (SL-BUP) induction period for all randomized subjects as well as the subjects who continued to study medication period (injectable formulation-experimental/ placebo) are reported here. Hence, the number of participants at risk is greater than the number started study medication in Participant flow module.
Arm/Group | Injectable Buprenorphine (BUP-inj) | Injectable Placebo (PBO-inj)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/13
Other Adverse Events (participants affected / at risk) | 4/5 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Injectable Buprenorphine (BUP-inj) (N=5) | Injectable Placebo (PBO-inj) (N=13)
Acute hypoxic and hypercapnic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Injectable Buprenorphine (BUP-inj) (N=5) | Injectable Placebo (PBO-inj) (N=13)
Adverse Drug Reaction (General disorders) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 4 (4)
Pain (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Electrocardiogram ST Segment elevation (Investigations) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Candida Infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 1 (1)
Tinnitis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Abscess Limb (Infections and infestations) | 0 (0) | 1 (1)
Chemical Burn on Skin (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urethritis (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal Gonococcal Infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT05283304/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT05283304/ICF_001.pdf